CLINICAL TRIAL: NCT02236026
Title: A Double-Blind, Placebo-Controlled, Randomized, Crossover Design Study With an Open-Label Active Control to Evaluate the Potential of Nestorone® to Delay Cardiac Repolarization in Healthy Female Volunteers: A Thorough QT/QTc Study
Brief Title: A Study With an Open-Label Active Control to Evaluate the Potential of Nestorone® to Delay Cardiac Repolarization in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 648
Record Dates: First submitted 2014-08-28; First posted 2014-09-10 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Nestorone use as an IV solution on heart rate;; Abnormality in Heart Rate or Rhythm, Unspecified as to Time of Onset
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Supratherapeutic dose of Nestorone (Experimental): Subjects will be randomized to a treatment sequence on Day 1 of Treatment Period 1, prior to administration of investigational product, according to a randomization schedule provided by the Sponsor
  Interventions: Drug: Supratherapuetic dose of Nestorone
- Placebo (Placebo Comparator): Subjects will be randomized to a treatment sequence on Day 1 of Treatment Period 1, prior to administration of investigational product, according to a randomization schedule provided by the Sponsor
  Interventions: Drug: Placebo
- Moxifloxacin (Experimental): Subjects will be randomized to a treatment sequence on Day 1 of Treatment Period 1, prior to administration of investigational product, according to a randomization schedule provided by the Sponsor
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Supratherapuetic dose of Nestorone
  Arms: Supratherapeutic dose of Nestorone
Drug: Placebo
  Arms: Placebo
Drug: Moxifloxacin
  Arms: Moxifloxacin

SUMMARY:
The purpose of the study is to evaluate the effect of Nestorone (NES) administered as an bolus injection on the corrected QT interval using Fridericia's formula (QTcF).

ELIGIBILITY:
Inclusion Criteria:

* Is a premenopausal female, ≥ 18 to < 40 years of age at the time of Screening;
* Has a BMI ≥ 18.5 and ≤ 32 kg/m2 (weight ≥ 50 kg) at Screening
* Is in a state of general good health based on medical history and physical examination;
* Is regularly menstruating (cycles of 22 to 35 days duration) over the previous 6 months prior to Screening, as reported by the subject;
* If of childbearing potential, must be practicing an acceptable non-hormonal, method of birth control until the end of the study (Exit/Early Termination). Such methods include but are not limited to: Sexual abstinence; Male or female condom in combination with spermicidal foam/gel/cream/ suppository; Vasectomized or female partner; Diaphragm/cervical cap with spermicide; Bilateral tubal ligation sterilization at least 6 months before the screening visit, or an ESSURE or ADIANA procedure with an hysterosalpingography confirmation test at least 6 months before the screening visit; Copper intrauterine device.
* Is able to fulfill the requirements of the protocol, and indicates a willingness to participate in the study by providing written informed consent and an authorization to disclose PHI.

Exclusion Criteria:

* Is pregnant or lactating;
* Has hypersensitivity or allergy to NES, moxifloxacin, or related compounds, or any of the inactive ingredients used in the investigational product formulations;
* Has a contraindication to progestin or estrogen therapy;
* Has impaired hypothalamic-pituitary-adrenal reserve, or history of oral glucocorticoid replacement therapy in 12 months prior to Screening.
* Has experienced undiagnosed genital bleeding, excluding inter-menstrual spotting, within 6 months of Screening;
* Has undergone a gynecological examination, which results in clinically significant abnormalities, at Screening;
* Has had treatment with oral, topical or vaginal steroid hormones (e.g., estrogens, progestogens, androgens [including dehydroepiandrosterone], corticosteroids) within 8 weeks prior to Screening, or treatment with injectable or implantable steroids at any time during the 6 months prior to Screening;
* Is currently using, or has used within 6 months prior to Screening, hormonal contraception or progestin intrauterine device.
* Has known or suspected carcinoma of the breast;
* Has benign or malignant liver tumors or acute liver disease;
* Has current or past thrombophlebitis or thromboembolic disorders or a family history of thromboembolic disorders;
* Has a personal history of myocardial disease, Long QT Syndrome or a personal or family history of Long QT Syndrome (e.g., Anderson-Tawil Syndrome [micrognathia, low set ears, clinodactyly]; Timothy's Syndrome [syndactyly and autism spectrum disorder];: Jervell/Lange-Nielsen Syndrome [bilateral hearing loss]; Romano-Ward Syndrome [fainting, seizures]), unexplained syncope or presyncope, or current or recurrent hypokalemia.
* Has a family history in genetically related grandparents, parents, uncles/aunts, cousins, or children of Long QT Syndrome, non-ischemic cardiomyopathy, or unexplained sudden death before 50 years of age.
* Has an abnormal 12-lead ECG, with clinically significant abnormalities of rate, rhythm, or conduction including: HR < 45 or > 90 beats per minute (bpm), after a 5 minute supine rest; PR interval > 220 ms; QRS interval > 120 ms; QTcF or corrected QT interval using Bazett's formula (to be determined by Investigator) > 450 ms; QTcF < 300 ms; Any degree of clinically significant fascicular block, bundle branch block, or intraventricular conduction delay; QRS and/or T wave that the Investigator judges to be unfavorable for consistently accurate QT measurements (e.g., indistinct QRS onset, low amplitude T wave, inverted or terminally inverted T wave, merged T/U waves, indistinct T wave offset, or prominent U wave that affects QT measurement); Neuromuscular artifact that cannot be readily eliminated;
* Has, on ECG, premature atrial or ventricular beats or other findings that in the Investigator's opinion represent clinically significant excessive HR variation;
* Has any clinically significant deviation from normal in any of the screening tests or initial exams that, in the opinion of the Investigator, might present a safety risk for participation or would confound analysis or interpretation of the study results;
* Has participated in a clinical study or used any investigational drug within the 60 days prior to Screening;
* Requires the use of medication, including over-the-counter products, or nutritional supplements, with the exception of aspirin, ibuprofen, and acetaminophen. Medications are not exclusionary if they are discontinued as described below; however, under no circumstance should medication be discontinued if doing so would place a subject at risk; Medications (including nutritional supplements) known to be moderate or potent inhibitor of cytochrome P450 (CYP) 3A4, or to prolong the QT/QTc interval, must be discontinued at least 21 days prior to study entry (Day -1 of Treatment Period 1); All other prescription medications must be discontinued at least 14 days prior to study entry (Day -1 of Treatment Period 1), unless in the opinion of the Investigator the concomitant use of such medication does not place the subject at risk and will not confound the collection, analysis, or interpretation of study data; Over-the-counter medications (including nutritional supplements) must be discontinued at least 7 days prior to study entry (Day -1 of Treatment Period 1);
* Foods or beverages containing alcohol, caffeine, xanthine, or grapefruit are not allowed within 48 hours of Day -1 of each treatment period.
* Has a positive hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) screen;
* Has a positive test for alcohol or drugs of abuse, or a history of known or suspected alcohol or drug abuse;
* Has used tobacco products within 6 months prior to Screening, or has a positive urine test for tobacco use;
* Has donated more than 400 mL of blood/plasma in the 60 days prior to Day -1 of Treatment Period 1;
* Is unable or unwilling to provide written informed consent or comply with the activities or instructions of the study;
* Is judged by the Investigator to be unsuitable for any reason.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Nestorone (NES) administered as an IV solution on the corrected QT interval using Fridericia's formula (QTcF). | Days 1, 2, 30, 31, 32, and 33
  Measurement of any changes from baseline in heart rhythm using an electrocardiogram at different time points after receiving NES as an IV solution

CONTACTS AND LOCATIONS:
Overall Officials: George W. Creasy, MD, Study Director — Population Council
Locations (1):
- Harbor Hospital, 3001 South Hanover Street, 7th Floor, Baltimore, Maryland, United States